CLINICAL TRIAL: NCT06057714
Title: Quantitation and Spatial Registration of Airways Dysfunction With Dynamic 19F MRI in Cystic Fibrosis
Status: Recruiting | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 20-1233; 5K23HL138257-03 (NIH)
Record Dates: First submitted 2023-09-18; First posted 2023-09-28 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Cystic Fibrosis; Ventilatory Defect
MeSH Terms: conditions — Cystic Fibrosis | interventions — perflutren

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: All subjects to receive inhaled perfluoropropane via standard Douglas bag at every visit (3-5 visits). They will breathe the gas for 5 breath hold cycles (variable volumes as lung capacity/size varies per participant). Not to exceed 30 liters inhaled at each visit as this is the max capacity of our Douglas bag.
  Interventions: Combination Product: 19F MRI

INTERVENTIONS:
Combination Product: 19F MRI — Inhalation of a biologically inert contrast gas, perfluoropropane, combined with 19F-tuned MRI with image acquisition at breath-hold and during tidal breathing
  Other Names: Perfluoropropane (PFP)

SUMMARY:
The purpose of this study is to look at lung ventilation in people with cystic fibrosis over time (1 year) using magnetic resonance imaging (MRI) with an inhaled contrast gas, and compare these measures to lung function assessed by spirometry and multiple breath nitrogen washout. This study also looks at how these measures change in response to a pulmonary exacerbation and treatment (if applicable). Over the span of a year, participants would be asked to complete 3-5 visits to the University of North Carolina at Chapel Hill (UNC). with each lasting up to 4 hours. If participants do not have a pulmonary exacerbation during the year they would be asked to complete 3 visits (one at enrollment, a second roughly 2 weeks later, and the third approximately a year later). If participants do experience a CF pulmonary exacerbation they would complete 5 visits (Visit 1, Visit 2, two exacerbation visits with one before treatment and the other after, and Visit 3 at one year after Visit 1). Only one exacerbation per participant will be tracked. Participants are eligible for this study if they are 18 years old or older, have Cystic Fibrosis (CF) with mild lung disease (FEV1 >/= 60%), and can undergo an MRI. There are no known benefits for participating in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be ≥18 years of age
2. Non-smokers (<10 pack/year history and no active smoking in the past year)
3. Diagnosis of cystic fibrosis via standard sweat chloride/phenotypic features/genotyping
4. No use of supplemental oxygen
5. Stable lung function (within 10% of personal best in the last 6 months) with no pulmonary exacerbations in the past 4 weeks and baseline FEV1≥60% of predicted
6. Evidence of a personally signed and dated consent indicating that the subject has been informed of all pertinent aspects of the trial
7. Subjects must be willing and able to comply with scheduled visits and other trial procedures

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the trial:

1. Active or past smokers or vapers with less than 1 year since quitting or >10 pack-year smoking history
2. Unable to undergo a 3.0-Tesla MRI exam of the lungs and chest because of contraindications including

   1. Occupation (past or present) of machinist, welder, or grinder;
   2. Injury to the eye involving a metallic object
   3. Injury to the body by a metallic object (bullet, bullet ball, shrapnel)
   4. Presence of a cardiac pacemaker or defibrillator
   5. Presence of aneurysm clips
   6. Presence of carotid artery vascular clamp
   7. Presence of neurostimulator
   8. Presence of insulin or infusion pump
   9. Presence of implanted drug infusion device that is not known to be MRI compatible (i.e., was placed outside of UNC or is older than 10 years)
   10. Bone growth or fusion simulator
   11. Presence of cochlear, otologic or ear implant
   12. Any type of prosthesis (eye, penile, etc.)
   13. Artificial limb or joint
   14. Non-removable electrodes (on body, head or brain)
   15. Intravascular stents, filters or coils
   16. Shunt (spinal or intraventricular)
   17. Swan-Ganz catheter
   18. Any implant held in place by a magnet
   19. Transdermal delivery system (e.g. Nitro)
   20. An intrauterine device or diaphragm that is not MRI compatible
   21. Tattooed makeup (eyeliner, lips, etc.) or tattoos covering >25% of body surface area
   22. Body piercings (must be removed before MRI)
   23. Any metal fragments
   24. Internal pacing wires
   25. Metal or wire mesh implants
   26. Hearing aid (remove before MRI) aa. Dentures (remove before MRI) bb. Claustrophobia
3. Unable to tolerate inhalation of gas mixture
4. Presence of facial hair that may interfere with the fit of the mask (and unwillingness to shave prior to each MRI)
5. Any changes in medications that may affect CF lung disease in the past 28 days, including any experimental therapies
6. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the subject inappropriate for entry into this trial.
7. Pregnancy; women of childbearing potential must have a confirmed negative urine pregnancy test on the day of the MR scan, prior to the MRI scan.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with cystic fibrosis and stable lung disease at the time of enrollment
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Ventilation Defect Parameter (VDP) over 14 days | Day 1 to Day 14
  VDP measured at Day 1 and Day 14, expressed as a percentage of total lung volume
Change in VDP over 365 days | Day 1 to Day 365 (+/- 30 days)
  Average of VDP measured at Day 1 and Day 14; subtracted from VDP at Day 365, expressed as a percentage of total lung volume
Change in FLVlongtau2 over 14 days | Day 1 to Day 14
  FLVlongtau2 measured at Day 1 and Day 14, expressed as a percentage of total lung volume
Change in FLVlongtau2 over 365 days | Day 1 to Day 365 (+/- 30 days)
  Average of FLVlongtau2 measured at Day 1 and Day 14; subtracted from FLVlongtau2 at Day 365, expressed as a percentage of total lung volume
Change in VDP occurring with a protocol-defined CF pulmonary exacerbation | Day 1 to Day 365 (+/- 30 days)
  Difference in VDP between baseline and exacerbation visit 1, expressed as a percentage of total lung volume.
Change in FLVlongtau2 occurring with a protocol-defined CF pulmonary exacerbation | Day 1 to Day 365 (+/- 30 days)
  Difference in FLVlongtau2 between baseline and exacerbation visit 1, expressed as a percentage of total lung volume.

SECONDARY OUTCOMES:
Change in MRI severity score over 365 days | Day 1 to Day 365 (+/- 30 days)
  Change in MRI severity score from baseline to Day 365.
Correlation of MRI severity score with VDP at baseline. | Day 1 to Day 14
  Baseline is a mean of the VDP scores from Day 1 and Day 14 (expressed as percentage of lung).
  Correlation of MRI scores with VDP and FLVlongtau2
Correlation of MRI severity score with FLVlongtau2 at baseline. | Day 1 to Day 14
  Baseline is a mean of the FLVlongtau2 scores from Day 1 and Day 14 (expressed as percentage of lung).
  Correlation of MRI scores with VDP and FLVlongtau2

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Goralski, MD, Principal Investigator — UNC Chapel Hill
Locations (1):
- Univeristy of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No